CLINICAL TRIAL: NCT05981287
Title: Comparison of Task-oriented Activity Based Neurodevelopmental Principles and Gross Motor Task Training on Balance, Trunk Control and Functional Mobility in Children With Cerebral Palsy.
Brief Title: Comparison of Task-oriented Activity Based Neurodevelopmental Principles and Gross Motor Task Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0720
Record Dates: First submitted 2023-01-04; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy
Keywords: Balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented activities based on NDT (TOA-NDT) principle and Conventional Physical Therapy (Experimental): The experimental group undergo conventional physical therapy and additional task-oriented activities based on NDT (TOT-NDT) principle 10 - 36 sessions in 5-8 weeks, 2 to 6 days per sessions.
  Interventions: Other: Task-oriented activities based on NDT (TOA-NDT) principle and Conventional Physical Therapy
- Gross motor task training and Conventional physical therapy (CPT) (Active Comparator): This group will receive conventional physical therapy and additional gross motor task training 10-36 sessions in 5-8 weeks, 2 to 6 days per sessions.
  Interventions: Other: Gross motor task training and Conventional physical therapy (CPT)

INTERVENTIONS:
Other: Task-oriented activities based on NDT (TOA-NDT) principle and Conventional Physical Therapy — This will be a randomized clinical trial. patients are divided into two groups. one of them will undergo task-oriented activities along with conventional physical therapy treatment, while the other will undergo gross motor task training along with conventional physical therapy treatment. Purpose is to determine that which of them has greater benefit in improving balance trunk control and functional mobility in children with cerebral palsy.
  Other Names: Comparison between task oriented activities and gross motor task training
  Arms: Task-oriented activities based on NDT (TOA-NDT) principle and Conventional Physical Therapy
Other: Gross motor task training and Conventional physical therapy (CPT) — This will be a randomized clinical trial. patients are divided into two groups. one of them will undergo task-oriented activities along with conventional physical therapy treatment, while the other will undergo gross motor task training along with conventional physical therapy treatment. Purpose is to determine that which of them has greater benefit in improving balance trunk control and functional mobility in children with cerebral palsy.
  Other Names: Comparison between task oriented activities and gross motor task training
  Arms: Gross motor task training and Conventional physical therapy (CPT)

SUMMARY:
This study aims to find the comparison of task oriented activity based neurodevelopmental principles and gross motor task training on balance, trunk control and functional mobility in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) being a non-progressive neurodevelopmental condition, is the leading cause of chronic disability in children, making them physically and mentally handicapped and socially unapproachable. The low tone of the torso also causes postural instability, lack of mobility, and muscle stiffness in the legs. Therapeutic intervention for children with cerebral palsy should be composed of goal directed, functional, and meaningful activities by considering the clinical type, degree of disability, cognitive level and interest of the child. The trunk being the central key point of the body, proximal trunk control is a prerequisite for distal limb movement control, balance, and functional mobility. Since children with cerebral palsy show damage not only in the function and an ability to accomplish tasks, but also in the quality of movement. The objective of this study will be to help clinicians regarding the effectiveness of task-oriented training and gross motor functional training for children with cerebral palsy.

This will be a Randomized Clinical Trial in which participants of age 5 - 12 years with cerebral palsy will be assigned randomly for the study. Population will be taken from Physical Therapy Department of Agile Rehabilitation Complex, Bahawalpur. After taking consent, demographics including age, gender and birth history etc. will be recorded. Questionnaires will be distributed among parents and their responses will be collected. Questionnaires for trunk impairment scale, postural assessment scale, pediatric balance scale and GMFM-88 will be used as tools of assessment. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 27.0.

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic cerebral palsy
* Both boys and girls
* Age 5 - 12 years old
* Able to follow verbal commands
* Having level I or II of GMFCS

Exclusion Criteria:

* Uncooperative
* On antiepileptic and anti-spastic medications
* Having visual or intellectual impairments
* Having hearing deficit
* With any cardiac anomalies affecting exercise tolerance
* Less than 6-month post-orthopedic surgery or post-botulinum toxin injections

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale - PBS | 2 months
  Pediatric balance scale is an outcome measurement tool used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Trunk Control Measurement Scale - TCMS | 2 months
  Trunk Control Measurement Scale is the clinical tool to measure trunk control in children with cerebral palsy. Control of muscles is necessary to maintain stability around the trunk.
Gross Motor Function Measure 88 - GMFM 88 | 2 months
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. There are two versions of the GMFM - the original 88-item measure (GMFM-88) and the more recent 66-item GMFM (GMFM-66). The scoring system of the GMFM is a four-point scale that consists of 66 items divided into five dimensions of gross motor function:(a) lying and rolling, (b) sitting, (c) crawling and kneeling, (d) standing, and (e) walking, running and jumping.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Aamna Hassan, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No